CLINICAL TRIAL: NCT05012683
Title: To Assess the Utility of the Point Partial in a Clinical Take-home Study of Partial Hand Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Point Designs (Industry)
Collaborators: University of Colorado, Denver (Other); Arm Dynamics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 299090
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Results first posted 2024-01-23 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Amputation; Traumatic, Hand

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- No Prosthesis, then Prosthesis (Experimental): Baseline outcome measurements will be performed without a prosthesis. Then subject will be fit with a prosthesis and outcome measurements will be performed at 3 different points in time: immediately post-fitting, ~30 days post-fitting, and ~60 days post-fitting.
  Interventions: Device: Point Partial

INTERVENTIONS:
Device: Point Partial — Patient is fit with Point Partial partial finger prosthetic system

SUMMARY:
This study will allow us to assess whether the Point Partial confers functional and psychological benefit to persons with partial finger amputations in an unconstrained environment. The use of the Point Partial outside of the laboratory will allow for a wider variety of uses and for a more realistic simulation of the product being used in the field. This well-controlled trial (without randomization of subjects) will produce the first Level II-1 medical evidence in our field of partial hand prosthetic design as described by the 1989 U.S. Preventive Services Task Force. Furthermore, this study will provide important data to support providers who are requesting reimbursement from payers.

ELIGIBILITY:
Inclusion Criteria:

* Partial finger amputees with partial absence of index and/or middle fingers and presence of thumb. Additional finger loss is acceptable if all other criterion are met.
* Fluent in English
* Individuals aged 18 or greater
* Patients may present with either fused or mobile MCP joints.

Exclusion Criteria:

* Significant cognitive deficits as determined upon clinical evaluation
* Significant neurological deficits as determined upon clinical evaluation
* Significant physical deficits of the residual limb impacting full participation in the study as determined upon clinical evaluation
* Uncontrolled pain or phantom pain impacting full participation in the study as determined upon OT evaluation
* Serious uncontrolled medical problems as judged by the project therapist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Point Designs, Lafayette, Colorado
  - Arm Dynamics, Overland Park, Kansas
  - Arm Dynamics, Maple Grove, Minnesota
  - Arm Dynamics, Portland, Oregon
  - Arm Dynamics, Philadelphia, Pennsylvania
  - Arm Dynamics, Houston, Texas
  - Arm Dynamics, Irving, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- No Prosthesis, Then Prosthesis: Baseline outcome measurements will be performed without a prosthesis. Then subject will be fit with a Point Partial partial finger prosthetic system and outcome measurements will be performed at 3 different points in time: immediately post-fitting, ~30 days post-fitting, and ~60 days post-fitting.
Period: No Prosthesis (Day 0)
Arm/Group | No Prosthesis, Then Prosthesis
Started | 11
Completed | 11
Not Completed | 0
Period: Prosthesis (Day 0)
Arm/Group | No Prosthesis, Then Prosthesis
Started | 11
Completed | 11
Not Completed | 0
Period: Prosthesis (Day 30)
Arm/Group | No Prosthesis, Then Prosthesis
Started | 11
Completed | 11
Not Completed | 0
Period: Prosthesis (Day 60)
Arm/Group | No Prosthesis, Then Prosthesis
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- No Prosthesis, Then Prosthesis: Baseline outcome measurements will be performed without a prosthesis
  Outcome measurements will be performed after the subject has been fit with a prosthesis at 3 different points in time: immediately post-fitting, ~30 days post-fitting, and ~60 days post-fitting
  Point Partial: Patient is fit with Point Partial partial finger prosthetic system
Arm/Group | No Prosthesis, Then Prosthesis
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Capacity Assessment of Prosthetic Performance for the Upper Limb (CAPPFUL)
Description: Capacity Assessment of Prosthetic Performance for the Upper Limb (CAPPFUL) provides a comprehensive, performance based measure for upper limb prosthetic use with any upper-limb functional prosthesis at any amputation level through assessment of commonplace activities that take place in various planes of movement. Scale Title: Overall Performance. Scale Minimum: 0. Scale Maximum: 100. Higher score indicates better outcome.
Time Frame: Day 0: no prosthesis (pre-fitting)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Prosthesis, Then Prosthesis
Number analyzed (Participants) | 11
score on a scale | 90.3 (5.1)

2. Primary Outcome: Disability of the Arm, Shoulder and Hand (DASH)
Description: The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale. Scale Title: DASH Score. Scale Minimum: 0. Scale Maximum: 100. Higher score indicates worse outcome.
Time Frame: Day 0: no prosthesis (pre-fitting)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Prosthesis, Then Prosthesis
Number analyzed (Participants) | 11
score on a scale | 34.5 (17.7)

3. Primary Outcome: EuroQol-5 Dimension (EQ-5D-5L)
Description: Descriptive system for health-related quality of life states in adults, consisting of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression), each of which has five severity levels that are described by statements appropriate to that dimension. Scale Title: EQ-5D-5L Score. Scale Minimum: 0. Scale Maximum: 100. Higher score indicates better outcome.
Time Frame: Day 0: no prosthesis (pre-fitting)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Prosthesis, Then Prosthesis
Number analyzed (Participants) | 11
score on a scale | 80.6 (12.1)

4. Primary Outcome: Capacity Assessment of Prosthetic Performance for the Upper Limb (CAPPFUL)
Description: as for outcome 1
Time Frame: Day 0: with prosthesis, immediately post-fitting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Prosthesis, Then Prosthesis
Number analyzed (Participants) | 11
score on a scale | 88.4 (7.9)

5. Primary Outcome: Disability of the Arm, Shoulder and Hand (DASH)
Description: as for outcome 2
Time Frame: Day 0: with prosthesis, immediately post-fitting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Prosthesis, Then Prosthesis
Number analyzed (Participants) | 11
score on a scale | 28.3 (16.3)

6. Primary Outcome: EuroQol-5 Dimension (EQ-5D-5L)
Description: as for outcome 3
Time Frame: Day 0: with prosthesis, immediately post-fitting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Prosthesis, Then Prosthesis
Number analyzed (Participants) | 11
score on a scale | 80.7 (11.5)

7. Primary Outcome: Capacity Assessment of Prosthetic Performance for the Upper Limb (CAPPFUL)
Description: as for outcome 1
Time Frame: ~Day 30: with prosthesis, 30 days post-fitting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Prosthesis, Then Prosthesis
Number analyzed (Participants) | 11
score on a scale | 91.7 (5.4)

8. Primary Outcome: Disability of the Arm, Shoulder and Hand (DASH)
Description: as for outcome 2
Time Frame: ~Day 30: with prosthesis, 30 days post-fitting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Prosthesis, Then Prosthesis
Number analyzed (Participants) | 11
score on a scale | 26.1 (12.5)

9. Primary Outcome: EuroQol-5 Dimension (EQ-5D-5L)
Description: as for outcome 3
Time Frame: ~Day 30: with prosthesis, 30 days post-fitting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Prosthesis, Then Prosthesis
Number analyzed (Participants) | 11
score on a scale | 81.9 (9.2)

10. Primary Outcome: Capacity Assessment of Prosthetic Performance for the Upper Limb (CAPPFUL)
Description: as for outcome 1
Time Frame: ~Day 60: with prosthesis, 60 days post-fitting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Prosthesis, Then Prosthesis
Number analyzed (Participants) | 11
score on a scale | 92.0 (7.3)

11. Primary Outcome: Disability of the Arm, Shoulder and Hand (DASH)
Description: as for outcome 2
Time Frame: ~Day 60: with prosthesis, 60 days post-fitting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Prosthesis, Then Prosthesis
Number analyzed (Participants) | 11
score on a scale | 19.0 (9.5)

12. Primary Outcome: EuroQol-5 Dimension (EQ-5D-5L)
Description: as for outcome 3
Time Frame: ~Day 60: with prosthesis, 60 days post-fitting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Prosthesis, Then Prosthesis
Number analyzed (Participants) | 11
score on a scale | 81.4 (16.8)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | No Prosthesis, Then Prosthesis
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT05012683/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT05012683/SAP_001.pdf